CLINICAL TRIAL: NCT01499745
Title: Exercise Training at Ambulatory Pulmonary Rehabilitation in Idiopathic Pulmonary Fibrosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Prof. Mordechai Kremer Head of Pulmonary Institute, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMCBH116531 CTIL
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis (IPF) patients
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training at Pulmonary Rehabilitation Program (Active Comparator): Exercise Training at Pulmonary Rehabilitation Program 2 weekly sessions of 60 min for 12 weeks
  Interventions: Behavioral: Pulmonary Rehabilitation
- Standard Treatment for IPF (Placebo Comparator): Continue for normal live with standard treatment
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — Exercise Training in Pulmonary Rehabilitation Program:
  12 weeks of 60 min exercise bout, twice a week at pulmonary rehabilitation

SUMMARY:
* Idiopathic pulmonary fibrosis (IPF) is a chronic progressive, fibrosing parenchymal lung disease with unknown etiology. The prevalence of IPF is estimated between 2-29 cases per 100,000 in general population with median survival rates of 2-5 years from time of diagnosed.
* Dyspnea and chronic dry cough are the prominent symptoms in those patients which cause to impaired functional capacity and quality of life (QOL).
* Drug therapy usually is ineffective approach, what makes a call for an effective treatment.
* Pulmonary Rehabilitation (PR) had been founded as safe and effective treatment in increasing functional capacity, decrease symptoms and improve QOL mainly among Chronic Obstructive Pulmonary Disease (COPD). However, recently growing evidence also supports the efficiency of PR in IPF patients.
* The Aim of the suggested study is to examine the effect of exercise training (ET) at ambulatory pulmonary rehabilitation among IPF patients.
* The investigators hypothesize that ET at PR program will increase functional capacity, will decrease level of dyspnea and improve QOL in IPF patients.
* Patients and Methods:
* 40 IPF patients males and females (aged 30-90 years old) will be recruiting to this study. After clinical assessment they will be randomly allocated to PR group n=20 or to Control group n=20.
* All patients will undergo a clinical assessment including medical history, risk factors for IPF and physical examination. On the first meeting at baseline and within one week post intervention (PR) the following measurements will be made: dyspnea score, QOL and physical activity level questionnaires. In addition, anthropometric measurements, echocardiography, blood samples, pulmonary function tests, cardiopulmonary exercise test, battery of functional test and 6 minute walk test (6MWT).
* The PR group will participate in 12 weeks of supervised group's ET program. The training program will be consisted two 6 week blocks of 60 min exercise bout twice a week. In the first block the patients will perform aerobic interval training with treadmill walking, cycling, and step climbing. In the second block, subjects will perform longer periods of continuous aerobic exercise, with resistance training by step climbing, unsupported arm/leg exercises with and without dumbbells (0.5-1 kg), and supporting body weight over a chair. Pulmonary function test and 6MWT will be also performed after completing first 6 week block. The control group will be assessed at baseline and after 12 weeks without participating in PR program.

ELIGIBILITY:
Inclusion Criteria:

* IPF patients diagnosed essentially according to the American Thoracic and European Respiratory Societies (ATS-ERS) by clinical diagnostic criteria of:
* High-resolution computed tomography (HRCT) demonstrating a pattern of "confident" or "possible" IPF (b) Abnormal pulmonary physiology with evidence of restriction and/or impaired gas exchange (can exist during exercise alone)
* Exclusion of other known causes of restrictive lung disease (e.g.: connective tissue disease, environmental exposure,etc

Exclusion Criteria:

* Patients with severe comorbid illnesses, unstable coronary artery disease, collagen vascular diseases and the need for high flow oxygen therapy (˃ 3-4 L\min).
* History of syncope on exertion or any comorbidities which precluded exercise training (such as severe orthopaedic or neurological deficits or unstable cardiac disease).
* Patients were also excluded if they had participated in a pulmonary rehabilitation program in the past 12 months.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | Before and after 12 weeks of Pulmonary Rehabilitation
  Peak oxygen consumption during standart cardiopulmonary exercise test on bicycle argometer
6 min walk test | Before and after 12 weeks of Pulmonary Rehabilitation
  distance covered in meters during 6 min of walking

SECONDARY OUTCOMES:
Echocardiography Parameters | Before and after 12 weeks of Pulmonary Rehabilitation
  Stroke Volume, Cardiac Output, Pulmonary Arterial Systolic Pressure
Blood tests | Before and after 12 weeks of Pulmonary Rehabilitation
  NT-proBNP, CRP
Medical Research Council (MRC) dyspnea score questionnaire | Before and after 12 weeks of Pulmonary Rehabilitation
St George's Respiratory Questionnaire (SGRQ) for evaluation quality of life | Before and after 12 weeks of Pulmonary Rehabilitation
International Physical Activity Questionnaire (IPAQ)- for estimation physical activity level | Before and after 12 weeks of Pulmonary Rehabilitation
Battery of 4 functional tests | Before and after 12 weeks of Pulmonary Rehabilitation
  1.30 seconds chair stand test- number of repetitions in 30 sec 2.Chair sit-and- reach test (trunk and hamstring flexibility) - number of cm on ruler 3.Back stretch (shoulder and back flexibility) - number of cm on ruler 4.8-ft-up-and -go (agility and coordination)- number of sec that takes to complete the task
Pulmonary function test | Before and after 12 weeks of Pulmonary Rehabilitation
  FVC, FEV1, FEV1\FVC, TLC, DLCO, FRC.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, M.D, Principal Investigator — Rabin Medical Center, Belinson Hospital
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Derived] Vainshelboim B, Kramer MR, Myers J, Unterman A, Izhakian S, Oliveira J. 8-Foot-Up-and-Go Test is Associated with Hospitalizations and Mortality in Idiopathic Pulmonary Fibrosis: A Prospective Pilot Study. Lung. 2019 Feb;197(1):81-88. doi: 10.1007/s00408-018-0189-4. Epub 2019 Jan 2. PMID 30600393
- [Derived] Vainshelboim B, Oliveira J, Fox BD, Kramer MR. The Prognostic Role of Ventilatory Inefficiency and Exercise Capacity in Idiopathic Pulmonary Fibrosis. Respir Care. 2016 Aug;61(8):1100-9. doi: 10.4187/respcare.04471. Epub 2016 May 10. PMID 27165419
- [Derived] Vainshelboim B, Fox BD, Kramer MR, Izhakian S, Gershman E, Oliveira J. Short-Term Improvement in Physical Activity and Body Composition After Supervised Exercise Training Program in Idiopathic Pulmonary Fibrosis. Arch Phys Med Rehabil. 2016 May;97(5):788-97. doi: 10.1016/j.apmr.2016.01.018. Epub 2016 Feb 8. PMID 26869288
- [Derived] Vainshelboim B, Oliveira J, Fox BD, Soreck Y, Fruchter O, Kramer MR. Long-term effects of a 12-week exercise training program on clinical outcomes in idiopathic pulmonary fibrosis. Lung. 2015 Jun;193(3):345-54. doi: 10.1007/s00408-015-9703-0. Epub 2015 Mar 3. PMID 25731736